CLINICAL TRIAL: NCT01357278
Title: Effect of Active Rehabilitation on Risk Factors for Fall, Bone Mineral Density, and the Quality of Life in Osteoporotic Patients. A Randomized, Controlled Intervention Study
Brief Title: Active Rehabilitation in Osteoporotic Patients
Acronym: ARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Kari Anne Hakestad, Kari Anne Hakestad, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: OsteoActive
Record Dates: First submitted 2010-04-21; First posted 2011-05-20 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Osteoporosis
Keywords: osteoporosis; exercise; intervention; rehabilitation; bone mineral density; muscle strength
MeSH Terms: conditions — Osteoporosis; Motor Activity | interventions — Rehabilitation; Patient Education as Topic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation and patient education (Experimental): Supervised rehabilitation consists of exercises for strength, balance and coordination twice weekly, and a home-training programme once weekly.
  Patient education will be offered every eight week.
  Interventions: Procedure: Rehabilitation and patient education
- Patient education (No Intervention): Patient education will be offered every eight week.

INTERVENTIONS:
Procedure: Rehabilitation and patient education — Supervised rehabilitation consists of exercises for strength, balance and coordination twice weekly, and a home-training programme once weekly.
  Patient education will be offered every eight week.
  Other Names: OsteoActive and OsteoInfo
  Arms: Rehabilitation and patient education

SUMMARY:
The main objective of this study is to target risk factors for falling, such as improved quadriceps muscle strength,balance and bone mineral density (BMD), to reduce the risk of osteoporotic fractures. Furthermore, to improve quality of life for patients with osteoporosis through an active rehabilitation program.

Sub-goals:

1. To assess the effect of active rehabilitation on risk factors for osteoporotic fractures (muscle strength, bone mineral density, balance and frequency of falling) in women with low bone mineral density (BMD)(t-score<1.5) and radius fracture?
2. To assess how active rehabilitation affect the quality of life of women with low bone mineral density(BMD) (t-score<1.5) and radius fracture?

DETAILED DESCRIPTION:
Norway has one of the worlds highest rates of fractures, and osteoporosis is a major risk factor. People with established osteoporosis (low bone density including fractures) experience a lot of pain, reduced physical function and quality of life. Treatments related to osteoporotic fractures cost the Norwegian society approximately five billion NOK per year. Over the past few years there has been an increasing focus on active rehabilitation in terms of physical activity as a major factor in preventing osteoporotic fractures. It is still unknown what type of training, as well as frequency, volume and intensity of activity that is necessary to achieve effect on risk factors for osteoporotic fractures. There are only limited organized exercise offers available for these patients, and health personals are quite often unsure what recommendations they should give. In addition, the patients are often hesitant participating in physical activities due to fear of falling and the risk of new fractures. The primary objective is therefore to assess if active rehabilitation can reduce the risk for osteoporotic fractures, as well as improving quality of life for women with established osteoporosis. The patients will be recruited from The Centre of Osteoporosis at Ulleval University Hospital and will be randomised into an intervention group (n=40) and a control group (n=40). The intervention consists of active rehabilitation 3 times a week for 6 months (OsteoActive). Our model is based upon the Canadian model. The results from the project will be published in international recognized scientific papers, and as information to health personals who work with this patient group. In the long term it is desirable that the clinicians treating osteoporotic patients can recommend active rehabilitation based upon a model developed on the findings from this study.

ELIGIBILITY:
Inclusion Criteria:

* Proven low bone mineral density (t-score < 1.5) plus radius fracture
* The radius fracture must not be older than 2 years, and must be healed by start of intervention (no plaster cast)
* Postmenopausal women above 50 years
* Domicile in the Oslo region

Exclusion Criteria:

* Hip fracture or vertebral fracture
* History of more than 3 osteoporotic fractures in different parts of the body
* Problems/illnesses indicating that active rehabilitation is not indicated
* Physical activity (moderate and hard intensity) for more than 4 hours a week
* Does not understand Norwegian, written and spoken

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Quadriceps Muscle Strength | Baseline
  Quadriceps muscle strength will be examined using isokinetic muscular strength tests on a Biodex machine (Biodex System 3 Pro, USA) and measured as peak torque (N-M) and total work of 60 and 180 degrees per second.
Quadriceps Muscle Strength | 6 months
  Quadriceps muscle strength will be examined using isokinetic muscular strength tests on a Biodex machine (Biodex System 3 Pro, USA) and measured as peak torque (N-M) and total work of 60 and 180 degrees per second.
Quadriceps Muscle Strength | 12 months
  Quadriceps muscle strength will be examined using isokinetic muscular strength tests on a Biodex machine (Biodex System 3 Pro, USA) and measured as peak torque (N-M) and total work of 60 and 180 degrees per second.

SECONDARY OUTCOMES:
Bone Mineral Density | Baseline
  Bone Mineral Density will be measured by means of "Double X-ray Absorptiometry" (DXA, Lunar, Prodigy). DXA is a measuring technique using x-rays with very low ray exposure. The method is exact, reliable, and the measuring time is briefer than for any other way to measure BMD. The scanned areas will be hip, femur neck and trochanter, arms, and lumbar spine.
Dynamic balance | Baseline
  Dynamic balance will be evaluated with Four Square Step Test (FSST).FSST is a dynamic standing balance test used to test balance in both multiple fallers (2 or more falls within the last 6 months) and non-multiple fallers (fewer than 2 falls within the last 6 months. Two FSST are completed using the best score of the two trials
The quality of life | Baseline
  The quality of life will be evaluated by means of SF-36. SF-36 measures the patient's own health related quality of life. The instrument is divided into eight sub-scales (physical function, role limitations, physical, bodily pain, general health, vitality, social function, role limitations, emotional, and mental health). The SF-36 is scored to a 0-100 scale for each sub-scale, the higher the score the better the health status.
Physical function/walking capacity | Baseline
  Physical function/walking capacity will be evaluated using the 6 minutes walk test. This test has been validated for measuring functional status in elderly people. Following the 6 minutes walk test, the subjects will answer the following question on "Borgsskala" for measuring how exhausting they experienced the walking test, "on a scale from 6-20, where 6 indicates very easy and 20 indicates very exhausting".
Physical activity level | Baseline
  Physical activity level will be registered using the validated self-reported level of physical activity for elderly, PASE.
Anthropometric data | Baseline
  Anthropometric data such as height, weight, absolute and percentage fat, plus fat-free mass, will be measured by means of weight- and height scales and DXA measurements.
Bone Mineral Density | 6 months
  Bone Mineral Density will be measured by means of "Double X-ray Absorptiometry" (DXA, Lunar, Prodigy). DXA is a measuring technique using x-rays with very low ray exposure. The method is exact, reliable, and the measuring time is briefer than for any other way to measure BMD. The scanned areas will be hip, femur neck and trochanter, arms, and lumbar spine.
Bone Mineral Density | 12 months
  Bone Mineral Density will be measured by means of "Double X-ray Absorptiometry" (DXA, Lunar, Prodigy). DXA is a measuring technique using x-rays with very low ray exposure. The method is exact, reliable, and the measuring time is briefer than for any other way to measure BMD. The scanned areas will be hip, femur neck and trochanter, arms, and lumbar spine.
Dynamic balance | 6 months
  Dynamic balance will be evaluated with Four Square Step Test (FSST).FSST is a dynamic standing balance test used to test balance in both multiple fallers (2 or more falls within the last 6 months) and non-multiple fallers (fewer than 2 falls within the last 6 months. Two FSST are completed using the best score of the two trials
Dynamic balance | 12 months
  Dynamic balance will be evaluated with Four Square Step Test (FSST).FSST is a dynamic standing balance test used to test balance in both multiple fallers (2 or more falls within the last 6 months) and non-multiple fallers (fewer than 2 falls within the last 6 months. Two FSST are completed using the best score of the two trials
The quality of life | 6 months
  The quality of life will be evaluated by means of SF-36. SF-36 measures the patient's own health related quality of life. The instrument is divided into eight sub-scales (physical function, role limitations, physical, bodily pain, general health, vitality, social function, role limitations, emotional, and mental health). The SF-36 is scored to a 0-100 scale for each sub-scale, the higher the score the better the health status.
The quality of life | 12 months
  The quality of life will be evaluated by means of SF-36. SF-36 measures the patient's own health related quality of life. The instrument is divided into eight sub-scales (physical function, role limitations, physical, bodily pain, general health, vitality, social function, role limitations, emotional, and mental health). The SF-36 is scored to a 0-100 scale for each sub-scale, the higher the score the better the health status.
Physical function/walking capacity | 6 months
  Physical function/walking capacity will be evaluated using the 6 minutes walk test. This test has been validated for measuring functional status in elderly people. Following the 6 minutes walk test, the subjects will answer the following question on "Borgsskala" for measuring how exhausting they experienced the walking test, "on a scale from 6-20, where 6 indicates very easy and 20 indicates very exhausting".
Physical function/walking capacity | 12 months
  Physical function/walking capacity will be evaluated using the 6 minutes walk test. This test has been validated for measuring functional status in elderly people. Following the 6 minutes walk test, the subjects will answer the following question on "Borgsskala" for measuring how exhausting they experienced the walking test, "on a scale from 6-20, where 6 indicates very easy and 20 indicates very exhausting".
Physical activity level | 6 months
  Physical activity level will be registered using the validated self-reported level of physical activity for elderly, PASE.
Physical activity level | 12 months
  Physical activity level will be registered using the validated self-reported level of physical activity for elderly, PASE.
Anthropometric data | 6 months
  Anthropometric data such as height, weight, absolute and percentage fat, plus fat-free mass, will be measured by means of weight- and height scales and DXA measurements.
Anthropometric data | 12 months
  Anthropometric data such as height, weight, absolute and percentage fat, plus fat-free mass, will be measured by means of weight- and height scales and DXA measurements.

CONTACTS AND LOCATIONS:
Overall Officials: May Arna Risberg, dr philos, Study Chair
Locations (1):
- NAR, Department of Orthopaedics, Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Hakestad KA, Torstveit MK, Nordsletten L, Risberg MA. Effect of exercises with weight vests and a patient education programme for women with osteopenia and a healed wrist fracture: a randomized, controlled trial of the OsteoACTIVE programme. BMC Musculoskelet Disord. 2015 Nov 14;16:352. doi: 10.1186/s12891-015-0811-z. PMID 26578370
- [Derived] Hakestad KA, Torstveit MK, Nordsletten L, Axelsson AC, Risberg MA. Exercises including weight vests and a patient education program for women with osteopenia: a feasibility study of the OsteoACTIVE rehabilitation program. J Orthop Sports Phys Ther. 2015 Feb;45(2):97-105, C1-4. doi: 10.2519/jospt.2015.4842. Epub 2015 Jan 10. PMID 25579693